CLINICAL TRIAL: NCT04121884
Title: Neurophysiological Mechanisms of Accelerated Resolution Therapy (ART)
Acronym: M-ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kevin Kip, Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00040159
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Depressive Symptoms; Stress Disorder, Acute; Prolonged Grief Disorder; Alcohol Abuse; Stress Disorders, Post-Traumatic
Keywords: Heart Rate Variability; Sleep; Electrocardiogram; Electroencephlogram; Alcohol Abuse; Prolonged Grief Disorder; Stress Disorder, Acute; Stress Disorders, Post-Traumatic; Depressive Symptoms; Power Spectral Density
MeSH Terms: conditions — Depression; Stress Disorders, Traumatic, Acute; Prolonged Grief Disorder; Alcoholism; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: A prospective, longitudinal, descriptive study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ART Treatment (Experimental): A broad patient representation of male and female adults; aged > 18 years; English speaking; and significant clinical symptoms of any of the following conditions: PTSD, Depression, ASD, Complicated Grief, and Alcohol Abuse.
  Interventions: Behavioral: Accelerated Resolution Therapy

INTERVENTIONS:
Behavioral: Accelerated Resolution Therapy — The ART protocol first uses the technique of imaginal exposure to elicit physiological reactions associated with patient recall from beginning to end (verbally or non-verbally) of a traumatic/distressing experience. As physiological reactions emerge, the participant is directed to focus their attention on the specific body-centric reactions while laterally performing smooth pursuit eye movements which are achieved by tracking the clinician's hand which oscillates from left-to-right at a short distance from the participant's eyes. Then the participant is directed to imagine a positive way in which they prefer to recall their experience(s), including emphasis on "replacing" negative images in the brain with positive images. This technique is based on the process of memory reconsolidation, which allows for "adding" of positive material to the recall of negative, highly emotional past experiences.
  Other Names: ART

SUMMARY:
In brief, ART is an innovative "mind-body" (body-centric) psychotherapy that makes use of established core components of trauma-focused therapy including imaginal exposure and imagery rescripting to promote memory reconsolidation, all facilitated as the patient is directed by the therapist to perform sets of lateral left-right eye movements similar to rapid eye movements (REM). The investigators propose to investigate how ART may directly influence heart rate variability (HRV), EEG power spectral densities, and sleep architecture in three aims. At the broadest level, the investigators postulate that both within individual ART sessions, and across the full course of treatment (e.g. up to 4 sessions), ART results in a profound shift from sympathetic (arousal) to parasympathetic (rest) nervous system balance, and that this shift can be reliably measured by neurophysiological assessment using electrocardiogram (ECG) and electroencephalogram (EEG) measurement.

DETAILED DESCRIPTION:
Our long-term goal is to understand, from a mechanistic perspective, how ART appears to result in rapid, successful treatment of PTSD and related comorbidities. This knowledge will help to identify target populations for treatment, and objective approaches in which to evaluate patient outcome response beyond conventional reliance on self-report measures. Thus, specific aims of our proposal, which will make use of wireless equipment for Electrocardiographic (ECG) measurement of Heart Rate Variability (HRV), and Electroencephalographic (EEG) measurements of power spectral densities and sleep architecture, are as follows:

1. To quantify and characterize changes in HRV, EEG power spectral densities, sleep architecture, and ANS balance within individual sessions of ART, as well as before and at the end of treatment with ART (up to 4 sessions).
2. To examine whether the aforementioned ART-induced changes in HRV, EEG power spectral densities, sleep architecture, and ANS balance vary substantially in the setting of primary treatment for symptoms of post- traumatic stress disorder (PTSD), depression, acute stress disorder, complicated grief, and/or alcohol abuse.
3. To assess the degree of concordance between ART-induced objective measurement of changes in HRV, EEG power spectral densities, sleep architecture, and ANS balance and self-report changes in symptoms of PTSD, depression, acute stress disorder, complicated grief, and/or alcohol abuse.

The investigators will accomplish these objectives using a prospective, longitudinal, descriptive design to achieve robust results. Subjects (n=40) will be enrolled in the study based on symptomatology. All subjects will receive Accelerated Resolution Therapy (ART) on a weekly basis for up to 4 sessions. The dose of up to 4 sessions has been selected to insure what is believed to be an effective dose based on previous studies of ART for treatment of PTSD. The investigators will collect data pre, during, and post each ART session. The sample of 40 subjects will be drawn from referrals at private practices of designated licensed mental health clinicians certified in ART, referrals from stakeholders and academic and community partners (e.g. USF student veterans referred through the USF Office of Student Veterans), and referrals of immediate family members of an individual who received hospice care prior to death at Suncoast Hospice or Chapters Health System. All subjects will undergo an intake assessment by a licensed clinical psychologist to determine study eligibility at USF.

The investigators expect to obtain support for our central hypothesis that ART modulates neurophysiological mechanisms through neurophysiological biomarkers of the autonomic (parasympathetic) nervous system and improved sleep architecture. Knowledge from a mechanistic perspective, on how ART appears to result in rapid, successful treatment of symptoms of PTSD and related conditions will help to identify target populations for treatment, and objective approaches in which to evaluate patient outcome response beyond conventional reliance on self-report measures.

ELIGIBILITY:
Inclusion Criteria:

* Posttraumatic Stress Disorder (PTSD): Score of > 33 on the 20-item DSM-V PTSD Checklist (PCL-V) or
* Depression: Score of > 16 on the 20-item Center for Epidemiologic Depression Scale or
* Acute stress disorder: Presence of criterions A-E on the 19-item Acute Stress Disorder Scale or
* Complicated grief: Score of > 25 on the 19-item Inventory of Complicated Grief or
* Alcohol abuse: Score of > 10 on 10-item Alcohol Use Disorders Identification Test (AUDIT) and
* Corroboration of the above symptomatology through verification of the corresponding subscale of the 125-item Psychiatric Diagnostic Screening Questionnaire (PDSQ).

Exclusion Criteria:

* Currently engaged in another psychotherapy regimen including currently engaged in ART or another eye movement therapy, such as EMDR;
* Have a major psychiatric disorder (e.g. bipolar disorder) deemed likely to interfere with treatment delivery;
* Currently in a formal substance dependence treatment program (alcohol and/or drug) anticipated to interfere with treatment delivery (e.g. through detox and symptoms of physiological withdrawal). All persons recruited for potential study participation will undergo a clinical intake assessment, with completion of ART intake form, by a licensed clinical therapist, to determine study eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Autonomic Nervous System (ANS) Imbalance | Baseline pre first ART session at study day 1 and post 4th ART session at 5 weeks
  HRV, EEG power spectral densities, and sleep architecture

SECONDARY OUTCOMES:
Changes in ANS During ART | During first ART session at 1 week and during 4th ART session at 5 weeks
  HRV and EEG power spectral densities

OTHER OUTCOMES:
Degree of concordance between ART-induced changes in ANS and symptoms of PTSD, depression, ASD, complicated grief, and alcohol abuse | Baseline pre first ART session at study day 1 and post 4th ART session at 5 weeks
  DSM-V PTSD Checklist (PCL-V)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Kip, PhD, Principal Investigator — University of South Florida; Paula L Cairns, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kip KE, Sullivan KL, Lengacher CA, Rosenzweig L, Hernandez DF, Kadel R, Kozel FA, Shuman A, Girling SA, Hardwick MJ, Diamond DM. Brief treatment of co-occurring post-traumatic stress and depressive symptoms by use of accelerated resolution therapy((R)). Front Psychiatry. 2013 Mar 8;4:11. doi: 10.3389/fpsyt.2013.00011. eCollection 2013. PMID 23482431
- [Background] Kip KE, Hernandez DF, Shuman A, Witt A, Diamond DM, Davis S, Kip R, Abhayakumar A, Wittenberg T, Girling SA, Witt S, Rosenzweig L. Comparison of Accelerated Resolution Therapy (ART) for Treatment of Symptoms of PTSD and Sexual Trauma Between Civilian and Military Adults. Mil Med. 2015 Sep;180(9):964-71. doi: 10.7205/MILMED-D-14-00307. PMID 26327548
- [Background] Kip KE, Diamond DM. Clinical, Empirical, and Theoretical Rationale for Selection of Accelerated Resolution Therapy for Treatment of Post-traumatic Stress Disorder in VA and DoD Facilities. Mil Med. 2018 Sep 1;183(9-10):e314-e321. doi: 10.1093/milmed/usy027. PMID 29635395
- [Background] Kip KE, D'Aoust RF, Hernandez DF, Girling SA, Cuttino B, Long MK, Rojas P, Wittenberg T, Abhayakumar A, Rosenzweig L. Evaluation of brief treatment of symptoms of psychological trauma among veterans residing in a homeless shelter by use of Accelerated Resolution Therapy. Nurs Outlook. 2016 Sep-Oct;64(5):411-23. doi: 10.1016/j.outlook.2016.04.006. Epub 2016 May 7. PMID 27601310
- [Background] Kip KE, Shuman A, Hernandez DF, Diamond DM, Rosenzweig L. Case report and theoretical description of accelerated resolution therapy (ART) for military-related post-traumatic stress disorder. Mil Med. 2014 Jan;179(1):31-7. doi: 10.7205/MILMED-D-13-00229. PMID 24402982
- [Background] Hernandez DF, Waits W, Calvio L, Byrne M. Practice comparisons between accelerated resolution therapy, eye movement desensitization and reprocessing and cognitive processing therapy with case examples. Nurse Educ Today. 2016 Dec;47:74-80. doi: 10.1016/j.nedt.2016.05.010. Epub 2016 May 21. PMID 27250615
- [Background] Kip KE, Rosenzweig L, Hernandez DF, Shuman A, Diamond DM, Girling SA, Sullivan KL, Wittenberg T, Witt AM, Lengacher CA, Anderson B, McMillan SC. Accelerated Resolution Therapy for treatment of pain secondary to symptoms of combat-related posttraumatic stress disorder. Eur J Psychotraumatol. 2014 May 7;5. doi: 10.3402/ejpt.v5.24066. eCollection 2014. PMID 24959325
- [Background] Schimmels J, Waits W. A Tale of Two Compulsions - Two Case Studies Using Accelerated Resolution Therapy (ART) for Obsessive Compulsive Disorder (OCD). Mil Med. 2019 May 1;184(5-6):e470-e474. doi: 10.1093/milmed/usy257. PMID 30295890
- [Background] Blechert J, Michael T, Grossman P, Lajtman M, Wilhelm FH. Autonomic and respiratory characteristics of posttraumatic stress disorder and panic disorder. Psychosom Med. 2007 Dec;69(9):935-43. doi: 10.1097/PSY.0b013e31815a8f6b. Epub 2007 Nov 8. PMID 17991823
- [Background] Chalmers JA, Quintana DS, Abbott MJ, Kemp AH. Anxiety Disorders are Associated with Reduced Heart Rate Variability: A Meta-Analysis. Front Psychiatry. 2014 Jul 11;5:80. doi: 10.3389/fpsyt.2014.00080. eCollection 2014. PMID 25071612
- [Background] Thayer JF, Yamamoto SS, Brosschot JF. The relationship of autonomic imbalance, heart rate variability and cardiovascular disease risk factors. Int J Cardiol. 2010 May 28;141(2):122-31. doi: 10.1016/j.ijcard.2009.09.543. Epub 2009 Nov 11. PMID 19910061
- [Background] Thayer JF, Ahs F, Fredrikson M, Sollers JJ 3rd, Wager TD. A meta-analysis of heart rate variability and neuroimaging studies: implications for heart rate variability as a marker of stress and health. Neurosci Biobehav Rev. 2012 Feb;36(2):747-56. doi: 10.1016/j.neubiorev.2011.11.009. Epub 2011 Dec 8. PMID 22178086
- [Background] Kemp AH, Griffiths K, Felmingham KL, Shankman SA, Drinkenburg W, Arns M, Clark CR, Bryant RA. Disorder specificity despite comorbidity: resting EEG alpha asymmetry in major depressive disorder and post-traumatic stress disorder. Biol Psychol. 2010 Oct;85(2):350-4. doi: 10.1016/j.biopsycho.2010.08.001. Epub 2010 Aug 11. PMID 20708650
- [Background] Lobo I, Portugal LC, Figueira I, Volchan E, David I, Garcia Pereira M, de Oliveira L. EEG correlates of the severity of posttraumatic stress symptoms: A systematic review of the dimensional PTSD literature. J Affect Disord. 2015 Sep 1;183:210-20. doi: 10.1016/j.jad.2015.05.015. Epub 2015 May 15. PMID 26025367
- [Background] Todder D, Levine J, Abujumah A, Mater M, Cohen H, Kaplan Z. The quantitative electroencephalogram and the low-resolution electrical tomographic analysis in posttraumatic stress disorder. Clin EEG Neurosci. 2012 Jan;43(1):48-53. doi: 10.1177/1550059411428716. PMID 22423551
- [Background] Lee SH, Yoon S, Kim JI, Jin SH, Chung CK. Functional connectivity of resting state EEG and symptom severity in patients with post-traumatic stress disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2014 Jun 3;51:51-7. doi: 10.1016/j.pnpbp.2014.01.008. Epub 2014 Jan 19. PMID 24447944
- [Background] Metzger LJ, Paige SR, Carson MA, Lasko NB, Paulus LA, Pitman RK, Orr SP. PTSD arousal and depression symptoms associated with increased right-sided parietal EEG asymmetry. J Abnorm Psychol. 2004 May;113(2):324-9. doi: 10.1037/0021-843X.113.2.324. PMID 15122952
- [Background] Harvey AG, Jones C, Schmidt DA. Sleep and posttraumatic stress disorder: a review. Clin Psychol Rev. 2003 May;23(3):377-407. doi: 10.1016/s0272-7358(03)00032-1. PMID 12729678
- [Background] Germain A. Sleep disturbances as the hallmark of PTSD: where are we now? Am J Psychiatry. 2013 Apr;170(4):372-82. doi: 10.1176/appi.ajp.2012.12040432. PMID 23223954
- [Background] Levendowski DJ, Popovic D, Berka C, Westbrook PR. Retrospective cross-validation of automated sleep staging using electroocular recording in patients with and without sleep disordered breathing. Int Arch Med. 2012 Jun 25;5(1):21. doi: 10.1186/1755-7682-5-21. PMID 22726270
- [Background] Stepnowsky C, Levendowski D, Popovic D, Ayappa I, Rapoport DM. Scoring accuracy of automated sleep staging from a bipolar electroocular recording compared to manual scoring by multiple raters. Sleep Med. 2013 Nov;14(11):1199-207. doi: 10.1016/j.sleep.2013.04.022. Epub 2013 Aug 16. PMID 24047533
- [Background] Modarres MH, Opel RA, Weymann KB, Lim MM. Strong correlation of novel sleep electroencephalography coherence markers with diagnosis and severity of posttraumatic stress disorder. Sci Rep. 2019 Mar 12;9(1):4247. doi: 10.1038/s41598-018-38102-4. PMID 30862872